CLINICAL TRIAL: NCT03564171
Title: A Randomized Controlled Feasibility Study Comparing a Multimodal Prehabilitation Protocol to Normal Care for Women Undergoing Neo-adjuvant Chemotherapy for Breast Cancer
Brief Title: Prehabilitation for Women Undergoing Pre-operative Chemotherapy for Breast Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Frances Wright, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 041-2018
Record Dates: First submitted 2018-03-18; First posted 2018-06-20 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer; Rehabilitation; Neoadjuvant Therapy; Feasibility Studies
MeSH Terms: conditions — Breast Neoplasms | interventions — Preoperative Exercise

STUDY DESIGN:
Intervention Model Description: 2 arms: Intervention and Control (chosen by closed envelope, 1:1 randomization)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Patients will receive standard treatment without added intervention.
- Intervention (Experimental): These patients will receive standard treatment plus multimodal intervention (prehabilitation program) including :
  exercise, nutritional counseling, stress counseling, smoking cessation) before starting chemotherapy.
  Interventions: Combination Product: Prehabilitation

INTERVENTIONS:
Combination Product: Prehabilitation — stress counseling, exercise, nutritional counseling, smoking cessation counseling
  Arms: Intervention

SUMMARY:
To assess recruitment rate, attrition, compliance with weekly exercise, smoking cessation, and quality of life with a multimodal prehabilitation protocol for women with breast cancer undergoing neo-adjuvant chemotherapy for breast cancer.

DETAILED DESCRIPTION:
Proposal: A randomized controlled feasibility study comparing a multi-modal prehabilitation protocol to usual care for women undergoing neo-adjuvant therapy for breast cancer.

Methods: Study population: Sixty patients who are undergoing curative intent neo-adjuvant chemotherapy for breast cancer will be randomized to intervention (n=30) or standard care (n=30) at a single site (Sunnybrook).

Intervention: A multi-modal program composed of an exercise prescription that will progressively increase in intensity and duration towards the current physical activity guidelines, nutritional counseling, stress counseling, and smoking cessation (as needed).

Intervention: Exercises will be instructed and demonstrated by a physiotherapist prior to the initiation of chemotherapy and will continue up until surgery. Nutritional and stress counseling, as well as smoking cessation, will be offered at initial consult with physiotherapist.

Exercise Protocol: The prehabilitation program entails a home-based exercise with both total-body physical exercise and exercises specific to the upper quadrant over the period between baseline assessment and surgery. The exercise prescription will be provided by a physiotherapist based upon the baseline assessment and will consist of a goal of 60 minutes of home-based, unsupervised exercise on 4 days per week, including aerobic and resistance training. Each session will be individualized and based upon the baseline assessment and generally include: a 5-minute warm-up, 25 minutes of moderate intensity aerobic exercise (for example: brisk walking, treadmill, stationary bike) (intensity of 3-6 on the 0-10 Rating of Perceived Exertion Scale) (attached, Appendix A) and 25 minutes of upper quadrant-specific training (Appendix B), and a 5-minute cool-down consisting of stretches (Appendix B). The program introduction will include a description and demonstration of all of the exercises that will follow the baseline assessment. The participant will have an opportunity to try the exercises in the presence of the physiotherapist who will provide corrective feedback if necessary. The physiotherapist will discuss safety precautions (posture, breathing, etc.) and provide the participant with an exercise manual that describes the exercises in the program and the safety precautions. To complete the exercises at home, each participant will be provided with resistance Theraband(s) (red and yellow) required to complete the upper quadrant exercises that they may keep at the end of the study. Training intensity progression will occur when the participant can complete the aerobic exercise with mild exertion and/or when the participant can complete 15 repetitions of a given upper quadrant exercise without eliciting at least moderate exertion (i.e. 3 to 6 on the Rating of Perceived Exertion scale). The prehabilitation program will be supported with a manual including institutionally created postoperative rehabilitation exercises that comprise a significant proportion of the preoperative exercise prescription. The physiotherapist will communicate with the participants every 2 weeks to ensure program compliance, support appropriate progression, and to address any barriers to exercise (including questions about appropriate exercise completion) that may prevent ongoing participation (see contact with team Table 1).

Grip Strength: Grip strength is commonly used to assess upper extremity strength in patients with breast cancer (Sagen 2009) and will be assessed via the "Jamar Hand" dynamometer according to established protocols.

Aerobic Fitness: Aerobic fitness will be measured using the 6-minute walk test (6 Minute Walk Test). This test is a practical standardized measure of functional capacity and has been widely used for measuring the submaximal level of functional capacity in cancer patients (Vardar 2015, Santa Mina 2014, Schmidt 2013). This test will measure the distance that the patient can walk on a flat, hard surface in a period of 6 minutes.

Nutrition counseling: The registered dietitian will provide an initial individualized nutrition assessment and counseling session. The consultation will be about 60 minutes in length and can be conducted in person or via telephone.

The patient's nutritional history, assessment of usual intake and weight history will be reviewed to help identify any nutritional issues/concerns. The session will focus on the goals of nutrition before and during treatment, provide strategies to help the patient optimize or enhance the nutritional quality of the diet, maintain a healthy weight and minimize weight gain and address any nutrition-related questions or concerns.

The registered dietitian will follow-up with the patient 4 weeks after the initial consultation to review the nutrition care goals and outcomes, answer questions re. any potential nutrition-related side effects from treatment and address any other questions or concerns.

The patient will be encouraged to contact the dietitian as needed during treatment for on-going support of if any nutrition related questions or concerns.

Stress counseling: Stress management intervention: Stress management intervention will consist of a 60-90 minute individual session with a psychiatrist specializing in psychosocial oncology. The therapy session will be cognitive-behavioral in orientation. The components will include a psychoeducational module on the stress response to physical symptoms; problem-solving and coping skills; relaxation techniques; and guided imagery. During the initial session, participants will be oriented conceptually to four types of interventions for reducing anxiety and coping with stress: (1) Progressive muscle relaxation; (2) mindfulness; (3) deep breathing; and (4) imagery/visualization. Each intervention will have accompanying written materials, which will also contain links to online audio materials. The additional materials contain written and spoken instructions allowing for self-directed learning and practice of each of the four stress-reducing interventions. Participants will be invited to choose one or two of the four strategies to practice with the therapist in the initial session, and in any subsequent sessions that participants attend. The therapist will instruct participants to choose one audio file to listen to at each chemotherapy session.

Optional face-to-face 60 minute individual booster sessions will be offered to participants on a monthly basis until surgery, in order to review problem solving and coping skills, relaxation techniques, and guided imagery. If patients are found to need a greater frequency of psychiatric intervention or undergo a psychiatric crisis, or if they require psychotropic medications at any point during the study, the PI will be informed and a referral will be made to an alternate psychiatrist (if the patient chooses) at the Odette Cancer Centre who is not involved in this study.

Every 2 weeks the patients in the intervention (prehabilitation arm) will be asked these questions:

At each telephone follow-up or email, the frequency of use and acceptability will be assessed with the following questions:

(1) Over the past two weeks, how often did you listen to one of the audio materials? Never Less than half the days More than half the days Once each day More than once per day

(2a) During your most recent chemotherapy session, did you listen to any of the audio materials? Yes; No (2b) If no, please explain why _______________

(3) In a general sense, how satisfied are you with the audio materials you have received? Very satisfied 5; Mostly satisfied 4; Indifferent 3; or mostly dissatisfied 2; Very dissatisfied 1

At the end of the prehabilitation sessions, patients will fill in an 'acceptability of psychotherapy' evaluation (CSQ scale).

Smoking cessation: If required. Sunnybrook has a comprehensive smoking cessation program in place. 16% of patients in the Odette Cancer Program are smokers (internal data). For those patients who identify as a smoker (answered "yes" to the question of "Have you used any forms of tobacco in the past 6 months?"), a brief smoking cessation intervention will be provided outlining the benefits of quitting as well as the impact of continued smoking on the treatments for cancer (chemotherapy, surgery and radiation). These patients will be given education on the use of nicotine replacement therapy and will be offered a redemption card for 4 boxes of free nicotine replacement therapy products of their choice and advised to speak with their pharmacist. Patients will also be encouraged to accept a referral to Smokers Helpline which provides free smoking cessation counseling (telephone, texting or web-based) with a Quit Coach.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older, able to give consent, ECOG 0-1

Exclusion Criteria:

* pregnant, > 80 years, medical contraindications to exercise. History of severe and persistent mental illness, cognitive impairment, recent suicide attempts or >11 on "Hospital Anxiety and Depression Scale". If very active (> 24) on the Godin-Shephard scale.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Recruitment rate (percent reported by the research analyst ) | 18 month
  What percent of eligible patients were successfuly recruitted in the study
Exercise compliance rate (percent reported by analysis of data) | 18 month
  number of exercise sessions per week and mean compliance rate (percent of the prescribed exercises within sessions)
Attrition rate (percent reported by data analysis) | 18 month
  what percent of the patients left the study?
Stress consultation compliance rate (percent reported by data analyst) | 18 months
  Percent of the patients that have satisfaction with counseling and use of education meterials that are provided to them.

SECONDARY OUTCOMES:
Quality of life (FACT-B questionnair) | 18 months
  The Functional Assessment of Cancer Therapy - Breast (FACT-B) is a validated quality of life scale for breast cancer survivors capturing subdomains of physical, social, emotional, and functional well-being as well as specific concerns for breast cancer. The FACT-An, a validated fatigue scale for cancer survivors, the PROMIS which looks at cognitive functioning will be used.
Physical activity volume | 6 months
  How much activity the patients complete on a weekly basis
Aerobic fitness (6 minute walk test) | 6 months
  How does 6 min walk test change after intervention and treatment in both arms.
Arm fitness (grip strength test) | 6 months
  Grip strength will be assessed and compared
Exercise tolerance ( FACT-An questionnair) | 6 months
  how the patients tolerate to the exercise program

CONTACTS AND LOCATIONS:
Overall Officials: Frances Wright, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No